CLINICAL TRIAL: NCT07322939
Title: Effects of Visual Indicator Exercises for the Trunk and Lower Extremities on Activity and Participation in Parkinson's Disease
Brief Title: Effects of Exercise With Visual Feedback in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Büşra Akıncı, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKU/Ph/1
Record Dates: First submitted 2025-12-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Balance Impairment; Exercise Training; Postural Control
Keywords: parkinson disease; balance; postural control; visual feedback; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard exercise program (Active Comparator): Participants in the standard exercise group will receive a physiotherapist-supervised exercise program, performed three times per week for a total duration of eight weeks.
  Interventions: Other: Control Group
- standard exercise program and visual feedback-based exercise program (Experimental): Participants in the standard exercise program and visual feedback-based exercise program group will receive a physiotherapist-supervised exercise program, performed three times per week for eight weeks.
  Interventions: Other: Control Group; Other: Visual Feedback Exercise Group

INTERVENTIONS:
Other: Control Group — The exercises will start with 6-8 repetitions and will increase by 2 repetitions each week. Cervical Region: Cervical rotation, lateral flexion, chin-tuck exercises Upper Extremity: Shoulder joint range of motion exercises with a wand, scapular adduction, shoulder retraction Lower Extremity: Bridge exercise, hip flexion, extension, abduction exercises, knee extension exercises, ankle dorsiflexion - plantar flexion exercises Balance Exercises: Perturbation exercises with eyes open and eyes closed on a hard surface, perturbation exercises with eyes open and eyes closed on a soft surface, maintaining a tandem stance Ambulation: Walking training on a treadmill with a Modified Borg Scale of level 3-4. Walking training will begin with 6 minutes in the first week and will increase by 1 minute each week.
Other: Visual Feedback Exercise Group — The visual feedback exercise will be performed using a wearable laser pointer attached to the trunk and lower extremities, along with a visual tracking screen. The exercise duration is 20 minutes. The laser placed on the trunk will be used in various exercises, including maintaining stability in a seated position, on a Swiss ball, while standing, during different movements, and on various surfaces. Additionally, trunk control exercises will involve rotational, vertical-horizontal, and circular movements. Exercises targeting trunk control in a crawling position will also be included. For the lower extremities, the program will focus on ankle dorsiflexion, hip abduction and extension, and knee extension. All exercises will be progressively individualized on a weekly basis.
  Arms: standard exercise program and visual feedback-based exercise program

SUMMARY:
Patients with Parkinson's disease who apply to the Hasan Kalyoncu University Application and Research Center and meet the inclusion criteria will be included in the study. The included participants will be randomly assigned into either the intervention group or the control group using a sealed-envelope method. Both groups will undergo a standard exercise program, consisting of posture, strengthening, and balance training, under the supervision of a physiotherapist for 8 weeks, 3 days per week. In addition to this, the intervention group will receive an additional exercise program incorporating visual feedback using a laser pointer, targeting the trunk and lower extremities, also under the supervision of a physiotherapist for 8 weeks, 3 days per week.

DETAILED DESCRIPTION:
This study aims to investigate the effects of visual feedback exercise training focused on balance, postural control, and lower extremity mobility using a laser pointer, in addition to standard rehabilitation, on activity and participation in individuals with Parkinson's disease.

Hypotheses:

H1: Incorporating visual feedback-based trunk and lower extremity exercises using a laser pointer into standard rehabilitation improves body structure and function in individuals with Parkinson's disease.

H2: Incorporating visual feedback-based trunk and lower extremity exercises using a laser pointer into standard rehabilitation enhances activity and participation in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria

* Individuals diagnosed with idiopathic Parkinson's disease
* Disease severity classified as stage 1 to 3 according to the Modified Hoehn and Yahr Scale
* Patients receiving oral antiparkinsonian treatment only

Exclusion Critera

* Presence of musculoskeletal, cardiovascular, or vestibular disorders that may interfere with the completion of the assessments or treatment protocol
* Presence of additional neurological or psychiatric disorders other than Parkinson's disease
* Presence of visual impairment insufficient to perceive visual feedback

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Center of Pressure Elliptical Area | up to 8 weeks
  Postural control will be assessed using the Gyko wearable device. After the wearable vest is properly fitted, the participant will be asked to maintain balance for 30 seconds under four conditions: firm surface with eyes open, firm surface with eyes closed, soft surface with eyes open, and soft surface with eyes closed.
  The elliptical area of center of pressure displacement (mm²) obtained from the Gyko system will be recorded for each condition and used as the primary outcome measure.
Berg Balance Scale | up to 8 weeks
  The Berg Balance Scale is used to assess functional balance. It evaluates both dynamic and static balance through 14 tasks related to different positions, postural changes, and mobility. Each task is scored between 0 and 4 based on the individual's ability to perform the task independently, for a certain period, or over a specific distance (0: unable to perform, 4: normal performance). The highest possible score on the scale is 56, and a higher score indicates greater independence.

SECONDARY OUTCOMES:
L Test | up to 8 weeks
  The L Test is a functional mobility assessment. The participant starts from a seated position in a chair without armrests and, upon command, walks at a comfortable speed to a marked 3-meter point, turns right, continues walking for 7 meters, turns around, and returns to sit in the chair. The total time to complete the test (seconds) will be recorded.
Unified Parkinson's Disease Rating Scale | up to 8 weeks
  The first section evaluates non-motor features, the second section assesses activities of daily living, the third section involves motor examination, and the fourth section evaluates treatment complications. The four sections total 42 items. Each item is scored from 0 (no symptoms or signs) to 4 (the most severe symptoms or signs).
New York Postural Assessment Test | up to 8 weeks
  For each of the 13 body segments, three diagrams are provided. The posterior view includes the head, shoulders, spine, hips, and feet, while the lateral view includes the neck, chest, shoulders, upper back, trunk, abdomen, and lumbar region. Each body segment is scored as follows: 5 points (correct posture), 3 points (moderate deviation), and 1 point (severe deviation). The total score ranges from 13 to 65. A higher score indicates better posture.
Visual Analog Scale | up to 8 weeks
  Pain intensity was assessed using the Visual Analog Scale (VAS), which consists of a 100-mm horizontal line with scores ranging from 0 to 100 mm. Participants were instructed to mark the point on the line that best represented their current pain intensity, where 0 indicated "no pain" and 100 indicated "worst imaginable pain." The distance in millimeters from the left end of the line to the marked point was measured using a ruler. Higher VAS scores indicate greater pain intensity.
Parkinson Fatigue Scale | up to 8 weeks
  Consists of a total of 16 questions related to fatigue. Participants are asked to rate their agreement with the statements on a scale from 1 to 5 (1: strongly disagree, 5: strongly agree). The test result is determined by calculating the average of the responses to all questions.
10-Meter Walk Test | up to 8 weeks
  Gait speed will be assessed using the 10-Meter Walk Test. Participants will be instructed to walk a marked 10-meter distance at their usual walking speed. The time taken to complete the distance will be recorded, and walking speed (m/s) will be calculated.
Activities-specific Balance Confidence Scale | up to 8 weeks
  It consists of 16 tasks related to daily living activities performed both indoors and outdoors. Each item is rated on a scale from 0% (no confidence) to 100% (full confidence). Scores below 67% indicate a risk of falling, while higher scores reflect greater balance confidence.
Functional Reach Test | up to 8 weeks
  Postural stability will be assessed using the Functional Reach Test. The participant stands next to a wall with the arm closest to the wall elevated to 90° of shoulder flexion. The initial and final positions of the third finger are marked, and the reach distance (cm) is calculated.
Five Times Sit-to-Stand Test | up to 8 weeks
  Lower extremity strength and functional mobility will be evaluated using the Five Times Sit-to-Stand Test. Participants are instructed to stand up and sit down five times as quickly as possible from an armless chair with arms crossed. The total completion time (seconds) is recorded.
Freezing of Gait Questionnaire | up to 8 weeks
  Used to assess freezing episodes in patients with Parkinson's disease. It consists of six questions, each scored on a 0 to 4 scale (0: no symptoms, 4: severe). The total score ranges from 0 to 24, with higher scores indicating more severe freezing-related impairment.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | up to 8 weeks
  İt consists of 39 items divided into eight domains. Participants respond based on their experiences over the past month. Each question is scored on a 0 to 4 scale (0: never, 1: rarely, 2: sometimes, 3: often, 4: always).
  To calculate the domain score, the total score of the questions within that domain is summed, divided by the maximum possible score for that domain, and multiplied by 100.
  The total PDQ-39 score is obtained by summing the eight domain scores and dividing by 8, providing an overall quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Akıncı, Principal Investigator — Hasan Kalyoncu University; Günseli Usgu, Assoc. Prof., Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim KI, Im SC, Kim K. Effects of trunk stabilization exercises using laser pointer visual feedback in patients with chronic stroke: A randomized controlled study. Technol Health Care. 2023;31(2):471-483. doi: 10.3233/THC-220100. PMID 36120797